CLINICAL TRIAL: NCT01316263
Title: A Phase 2 Study of a Human Anti-PDGFRα Monoclonal Antibody (IMC-3G3) in Previously Treated Patients With Unresectable and/or Metastatic Gastrointestinal Stromal Tumors (GIST)
Brief Title: A Study of Olaratumab (IMC-3G3) in Previously Treated Participants With Unresectable and/or Metastatic Gastrointestinal Stromal Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial terminated strategically due to poor accrual.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14244; CP15-1008 (Other: ImClone, LLC); I5B-IE-JGDH (Other: Eli Lilly and Company); 2010-022560-12 (EudraCT Number)
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — olaratumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PDGFRα mutation negative (Experimental): Participants with GIST with genotypes that do not have a PDGFRα mutation given 20 milligrams per kilogram (mg/kg) Olaratumab intravenously (IV) every 14 days.
  Interventions: Biological: Olaratumab
- PDGFRα mutation positive (Experimental): Participants with GIST with genotypes that have a PDGFRα mutation given 20 mg/kg Olaratumab IV every 14 days.
  Interventions: Biological: Olaratumab

INTERVENTIONS:
Biological: Olaratumab — Administered IV
  Other Names: LY3012207; IMC-3G3

SUMMARY:
The purpose of this study is to evaluate the tumor response of stable disease (SD), partial response (PR), or complete response (CR) [according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v1.1 criteria)] at 12 weeks in participants with Gastrointestinal Stromal Tumors (GIST) harboring platelet-derived growth factor receptor alpha (PDGFRα) mutations and patients with GIST not harboring PDGFRα mutations.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically or cytologically confirmed, unresectable and/or metastatic GIST
* Participant has measurable disease
* Participant has documented objective progression following, or intolerance to, treatment with both imatinib and sunitinib
* Participant's Eastern Cooperative Oncology Group (ECOG) performance status (PS) is 0 to 2
* Participant has either:

  1. prior results from growth factor receptor associated with tyrosine kinase activity (KIT) and PDGFRα mutation analysis that meet analytical criteria as defined for the on-study analysis of these mutations and tumor tissue (from either primary or metastatic tumor) that can be submitted for analysis within 30 days after the first dose of study therapy; or
  2. if prior results from KIT and PDGFRα mutation analysis are not available or do not meet analytical criteria as above, then tumor tissue (from either primary or metastatic tumor) must be submitted for genotype testing at the latest 28 days prior to the first dose of study therapy
* Participant has adequate hematologic, hepatic, renal and coagulation function
* Women of childbearing potential and sexually active males must agree to use adequate contraception prior to study and for at least 12 weeks after the last dose of IMC-3G3
* Participant has a life expectancy of ≥ 3 months

Exclusion Criteria:

* Participant has untreated central nervous system metastases, and as a result, is clinically unstable with regard to neurologic function
* Participant has a history of another primary cancer
* Participant has received any investigational therapy within 14 days prior to registration, or is currently enrolled in any other type of medical research
* Participant is receiving concurrent treatment with other anticancer therapy
* Participant has known human immunodeficiency virus (HIV) infection
* Participant has undergone major surgery within 28 days prior to registration
* If female, participant is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (2):
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Boston, Massachusetts
- Belgium (2):
  - ImClone Investigational Site, Edegem
  - ImClone Investigational Site, Leuven
- Germany (5):
  - ImClone Investigational Site, Bad Saarow
  - ImClone Investigational Site, Berlin
  - ImClone Investigational Site, Essen
  - ImClone Investigational Site, Mannheim
  - ImClone Investigational Site, Tübingen
- ImClone Investigational Site, Leiden, Netherlands
- ImClone Investigational Site, Warsaw, Poland
- ImClone Investigational Site, Madrid, Spain

REFERENCES:
- [Derived] Wagner AJ, Kindler H, Gelderblom H, Schoffski P, Bauer S, Hohenberger P, Kopp HG, Lopez-Martin JA, Peeters M, Reichardt P, Qin A, Nippgen J, Ilaria RL, Rutkowski P. A phase II study of a human anti-PDGFRalpha monoclonal antibody (olaratumab, IMC-3G3) in previously treated patients with metastatic gastrointestinal stromal tumors. Ann Oncol. 2017 Mar 1;28(3):541-546. doi: 10.1093/annonc/mdw659. PMID 28426120

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were considered to have completed Stage 1 of the study discontinued due to progressive disease (PD) or died.
Groups:
- PDGFRα Mutation Positive: 20 milligrams per kilogram (mg/kg) of Olaratumab (IMC-3G3) was administered intravenously (IV) on Day 1 of each cycle (14-day cycles) to participants with gastrointestinal stromal tumors (GIST) with genotypes that had a platelet-derived growth factor receptor alpha (PDGFRα) mutation.
- PDGFRα Mutation Negative (Wild-Type): 20 mg/kg of Olaratumab (IMC-3G3) was administered IV on Day 1 of each cycle (14-day cycles) to participants with GIST with genotypes that did not have a PDGFRα mutation.
Period: Overall Study
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Started | 7 | 14
Received Any Study Drug | 7 | 14
Completed | 7 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received any study drug.
Groups:
- PDGFRα Mutation Positive: 20 mg/kg of Olaratumab (IMC-3G3) was administered IV on Day 1 of each cycle (14-day cycles) to participants with GIST with genotypes that had a PDGFRα mutation.
- Total: Total of all reporting groups
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type) | Total
Number analyzed (Participants) | 7 | 14 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (7.90) | 48.9 (9.11) | 54.2 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 14 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 14 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5
  Spain | 0 | 1 | 1
  Poland | 2 | 4 | 6
  Belgium | 1 | 2 | 3
  Netherlands | 0 | 2 | 2
  Germany | 2 | 2 | 4
Eastern Cooperative Oncology Group Performance Status(ECOG PS) [Number; unit: participants] — ECOG classifies participants according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  0=Fully active, able to carry on all pre-disease performance without restriction; 1=Ambulatory, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2=Ambulatory, no work activities; 3=Partially confined to bed, limited self-care; 4=Completely disabled.
  participants
    ECOG PS =0 | 2 | 5 | 7
    ECOG PS =1 | 4 | 9 | 13
    ECOG PS ≥2 | 1 | 0 | 1
Type of Cancer-Gastrointestinal Stromal Tumor [Number; unit: participants] | 7 | 14 | 21
Histology-Cell Type [Number; unit: participants]
  Epitheloid Cell | 6 | 0 | 6
  Spindle Cell | 0 | 9 | 9
  Mixed/Combined | 0 | 4 | 4
  Other-unspecified | 1 | 1 | 2
Initial T Classification Staging at Diagnosis [Number; unit: participants] — Staging: T0=no evidence of primary tumor; Tis=Carcinoma in situ; T1 to 4=presence of tumors, higher numbers indicate increased size, extent or degree of penetration; TX=primary tumor could not be assessed.
  participants
    Tis | 0 | 1 | 1
    T2 | 1 | 3 | 4
    T3 | 0 | 4 | 4
    T4 | 3 | 1 | 4
    TX | 1 | 4 | 5
    Missing | 2 | 1 | 3
Initial N Classification Staging at Diagnosis [Number; unit: participants] — Staging: N0=no regional lymph nodes metastasis; N1 to N3=Regional lymph node metastasis, higher number indicated greater involvement.
  participants
    N0 | 5 | 11 | 16
    N1 | 0 | 1 | 1
    Missing | 2 | 2 | 4
Initial M Stage at Diagnosis [Number; unit: participants] — Staging: presence or absence of distance metastasis, including lymph nodes that were not regional. M0=no distant metastasis; M1=distant metastasis; MX=distance metastasis could not be assessed.
  participants
    M0 | 4 | 7 | 11
    M1 | 1 | 5 | 6
    MX | 0 | 1 | 1
    Missing | 2 | 1 | 3
Current T Classification Staging [Number; unit: participants] — Staging: T0=no evidence of primary tumor; Tis=Carcinoma in situ; T1 to 4=presence of tumors, higher numbers indicate increased size, extent or degree of penetration; TX=primary tumor could not be assessed.
  participants
    T0 | 2 | 2 | 4
    T3 | 0 | 4 | 4
    T4 | 2 | 2 | 4
    TX | 2 | 4 | 6
    Unknown | 0 | 1 | 1
    Missing | 1 | 1 | 2
Current N Classification Staging [Number; unit: participants] — Staging: N0=no regional lymph nodes metastasis; N1 to N3=Regional lymph node metastasis, higher number indicated greater involvement.
  participants
    N0 | 5 | 8 | 13
    N1 | 0 | 3 | 3
    N2 | 1 | 0 | 1
    Missing | 1 | 3 | 4
Current M Classification Staging [Number; unit: participants] — Staging: presence or absence of distance metastasis, including lymph nodes that were not regional. M0=no distant metastasis; M1=distant metastasis; MX=distance metastasis could not be assessed.
  participants
    M1 | 6 | 13 | 19
    Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Tumor Response of Stable Disease (SD), Partial Response (PR) or Complete Response (CR) (Clinical Benefit Rate) at 12 Weeks
Description: Clinical benefit was defined as CR, PR, or SD using Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST, v1.1) criteria. CR: disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 millimeters (mm). PR: ≥30% decrease in sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter. SD: neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started. PD: increase ≥20% in sum of the diameters of target lesions, taking as reference the smallest sum on study (included baseline sum if that was the smallest on study). Sum must also have demonstrated an absolute increase of ≥5 mm, or appearance of 1 or more new lesions was considered progression. Percentage of participants=(participants with CR+PR+SD/participants in group) *100.
Time Frame: 12 weeks
Population: All participants who received any study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Number analyzed (Participants) | 7 | 14
percentage of participants | 42.9 [12.9 to 77.5] | 14.3 [2.6 to 38.5]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS defined as the duration from date of first dose of study drug until first radiographic documentation of PD using RECIST, v1.1 criteria or death from any cause. PD defined as ≥20% increase in the sum of diameters of target lesions, taking as reference smallest sum on study (included baseline sum if that was the smallest on study); sum must have demonstrated an absolute increase of ≥5 mm and the appearance of ≥1 new lesions was progression. Participants who died with no prior PD were considered to have progressed on day of death. Participants who did not progress or were lost to follow-up were censored at date of last radiographic tumor assessment; if no assessment was available censoring was at date of registration. If death or PD occurred after 2 consecutive missing radiographic visits censoring was date of last radiographic visit prior to missed visits. Use of new anticancer therapy prior to PD, censoring was date of last radiographic assessment prior to new therapy.
Time Frame: Baseline to the first date of objectively determined PD or death from any cause up to 35.9 weeks
Population: All participants who received any study drug. Censored participants: PDGFRα Mutant=2, PDGFRα Wild-Type=0.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Number analyzed (Participants) | 7 | 14
weeks | 32.1 [5.0 to 35.9] | 6.1 [5.7 to 6.3]

3. Secondary Outcome: Percentage of Participants With CR or PR [Radiographic Objective Response Rate (ORR)]
Description: The ORR was the best overall response of CR and PR using RECIST, v1.1 criteria. Participants who did not have a tumor response assessment for any reason were considered nonresponders and were included in the denominator that calculated the response rate. Percentage of participants = (number of participants achieving a response/total of participants treated) * 100.
Time Frame: Baseline up to 35.9 weeks and post study discontinuation 30-day follow-up
Population: All participants who received any study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Number analyzed (Participants) | 7 | 14
percentage of participants | 0 [NA to NA] — No participant achieved CR or PR. | 0 [NA to NA] — No participant achieved CR or PR.

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose of study drug to the date of death from any cause. Participants who were alive at the end of the post-study follow-up or were lost to follow-up were censored on the last date the participant was known to be alive.
Time Frame: Date of first dose of study drug to the date of death from any cause up to 57.3 weeks
Population: All participants who received any study drug. Participants censored: PDGFRα Mutant=4, PDGFRα Wild-type=4.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Number analyzed (Participants) | 7 | 14
weeks | NA [10.9 to NA] — Median and 90% Confidence Interval upper limit were not evaluable due to high number of censored participants. | 24.9 [14.4 to 49.1]

5. Secondary Outcome: Number of Participants With Adverse Events (AE) and Participants Who Died
Description: Clinically significant events were defined as serious AEs (SAEs) and other non-serious AEs, regardless of causality. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module. The number of participants who died due to an AE or disease progression are also reported.
Time Frame: Baseline up to 57.3 weeks and 30-day post study-discontinuation follow-up
Population: All participants who received any study drug.
Measure: Number; unit: participants
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Number analyzed (Participants) | 7 | 14
participants
  SAEs | 2 | 3
  AEs | 7 | 13
  Died Due to AE | 0 | 1
  Died Due to Disease Progression | 0 | 1

6. Secondary Outcome: Percentage of Participants With CR, PR or SD [Disease Control Rate (DCR)]
Description: DCR defined as CR, PR or SD using RECIST v1.1 criteria. CR was defined as the disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 mm. PR was defined as ≥30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify PD, taking as reference the smallest sum diameter since the treatment started. PD defined as ≥20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). Sum must also have demonstrated an absolute increase of ≥5 mm, or the appearance of 1 or more new lesions was considered progression. Percentage of participants=(number of participants with CR+PR+SD/number of participants in group) * 100.
Time Frame: Baseline up to 35.9 weeks
Population: All participants who received any study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Number analyzed (Participants) | 7 | 14
percentage of participants | 71.4 [34.1 to 94.7] | 28.6 [10.4 to 54.0]

7. Secondary Outcome: Maximum Concentration (Cmax)
Time Frame: Day 1 of Cycles 1 and 3 (14-day cycles)
Population: All participants who had evaluable pharmacokinetic (PK) Cmax results at the specific time point. Due to the limited data, Cmax is not representative of the study population.
Measure: Mean (Full Range); unit: nanograms per milliliter (ng/mL)
Groups:
- Olaratumab (IMC-3G3): 20 mg/kg of Olaratumab (IMC-3G3) was administered IV on Day 1 of each cycle (14-day cycles) to participants with GIST with genotypes that had a PDGFRα mutation or PDGFRα wild type.
Arm/Group | Olaratumab (IMC-3G3)
Number analyzed (Participants) | 3
nanograms per milliliter (ng/mL)
  Day 1 Cycle 1 (n=2) | 392.9 [314.0 to 471.8]
  Day 1 Cycle 3 (n=1) | 483.9 [NA to NA] — Individual values are reported when n <2.

8. Secondary Outcome: Area Under the Curve (AUC)
Time Frame: Day 1 of Cycles 1 and 3 (14-day cycles)
Population: Zero participants were analyzed. AUC was not reported. AUC could not be calculated due to an insufficient number of olaratumab serum concentrations.
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Half Life (t½)
Time Frame: Day 1 of Cycles 1 and 3 (14-day cycles)
Population: Zero participants were analyzed. t1/2 was not reported. t1/2 could not be calculated due to an insufficient number of olaratumab serum concentrations.
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Clearance (CL)
Time Frame: Day 1 of Cycles 1 and 3 (14-day cycles)
Population: Zero participants were analyzed. CL was not reported. CL could not be calculated due to an insufficient number of olaratumab serum concentrations.
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Time Frame: Day 1 of Cycles 1 and 3 (14-day cycles)
Population: Zero participants were analyzed. Vss was not reported. Vss could not be calculated due to an insufficient number of olaratumab serum concentrations.
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Participants With Human Anti-Olaratumab (IMC-3G3) Antibody Results
Description: Participants with Treatment Emergent (TE) anti-olaratumab (IMC-3G3) antibodies were participants with a 4-fold increase (2 dilutions) increase over a positive baseline antibody titer or for a negative baseline titer, a participant with an increase from the baseline to a level of 1:20.
Time Frame: Day 1 of Cycles 1, 3, 6, 12 and 18 prior to infusion (14-day cycles)
Population: All participants who received at least one dose of study drug and had evaluable baseline and evaluable post-baseline antibody data.
Measure: Number; unit: percentage of participants
Groups:
- PDGFRα Mutation Positive and Negative (Wild-Type): 20 mg/kg of Olaratumab (IMC-3G3) was administered IV on Day 1 of each cycle (14-day cycles) to participants with GIST with genotypes that had a PDGFRα mutation and that did not have a PDGFRα mutation.
Arm/Group | PDGFRα Mutation Positive and Negative (Wild-Type)
Number analyzed (Participants) | 19
percentage of participants | 5.3

ADVERSE EVENTS:
Arm/Group | PDGFRα Mutation Positive | PDGFRα Mutation Negative (Wild-Type)
Serious Adverse Events (participants affected / at risk) | 2/7 | 3/14
Other Adverse Events (participants affected / at risk) | 7/7 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDGFRα Mutation Positive (N=7) | PDGFRα Mutation Negative (Wild-Type) (N=14)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDGFRα Mutation Positive (N=7) | PDGFRα Mutation Negative (Wild-Type) (N=14)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Conjunctival pallor (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (9)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (5)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (6) | 5 (7)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (3) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood albumin increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 1 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (2)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Haematocrit increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Red blood cell count increased (Investigations) | 0 (0) | 1 (1)
Waist circumference increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (6)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Tearfulness (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The development of olaratumab (IMC-3G3) was put on hold in this indication due to reasons not related to efficacy and/or safety, Stage 2 of this study was not completed and trial terminated due to poor accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.